CLINICAL TRIAL: NCT05998291
Title: Gluteenittomaan Ruokavaliohoitoon Vastaamaton Ihokeliakia
Brief Title: Dermatitis Herpetiformis Refractory to Gluten Free Diet
Status: Enrolling by invitation | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other); University of Helsinki (Other)
Responsible Party: Sponsor
Other Study IDs: R23003
Record Dates: First submitted 2023-03-02; First posted 2023-08-18 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Dermatitis Herpetiformis
Keywords: dermatitis herpetiformis, dapsone, gluten-free diet
MeSH Terms: conditions — Dermatitis Herpetiformis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Refractory dermatitis herpetiformis patients: Dermatitis herpetiformis rash not controlled by strict glute-free diet
  Interventions: Other: Assessment of prognosis of refractory dermatitis herpetiformis. No intervention
- Dermatitis herpetiformis patients with good response to gluten-free diet: Dermatitis herpetiformis rash controlled by strict glute-free diet
  Interventions: Other: Assessment of prognosis of refractory dermatitis herpetiformis. No intervention

INTERVENTIONS:
Other: Assessment of prognosis of refractory dermatitis herpetiformis. No intervention — Assessment of prognosis of refractory dermatitis herpetiformis. No intervention

SUMMARY:
The main purpose of the study is to find out

1. the natural course of refractory dermatitis herpetiformis and the development of possible complications
2. the strictness of gluten-free diet treatment in refractory dermatitis herpetiformis

DETAILED DESCRIPTION:
Refractory dermatitis herpetiformis refers to dermatitis herpetiformis unresponsive to gluten-free diet therapy. So far, there is very little knowledge on the course of the disease and the causes and prognosis of refractory celiac disease.

Study patients with refractory dermatitis herpetiformis will be recruited. As a control material dermatitis herpetiformis patients with good response to gluten-free dietary treatment will be recruited.

ELIGIBILITY:
Inclusion Criteria:

Study patients:

* Dermatitis herpetiformis diagnosis
* Dermatitis herpetiformis rash not responding to a strict gluten-free diet after at least 3 years

Control patients:

* Dermatitis herpetiformis diagnosis
* Dermatitis herpetiformis with good response to a gluten-free diet

Exclusion Criteria:

Study patients:

-Not following strict gluten-free diet

Control patients:

-Not following a strict gluten-free diet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with refractory dermatitis herpetiformis
Sampling Method: Non-Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical prognosis | Baseline
  Occurrence of complications

SECONDARY OUTCOMES:
Dietary adherence GIP test, CDAT, TG2, TG3 and Ema antibodies, anamnesis | Baseline
  The strictness of gluten-free diet (GIP test)

OTHER OUTCOMES:
Microbiata | Baseline
  skin, oral and intestinal microbiata
Quality of life measure DLQI | Baseline
  DLQI (10-items, a higher score indicating lower quality of life)
Quality of life measure BGWP | Baseline
  PGWP (22-items with values 1-6, total score range 22-132, a higher score indicating better quality of life)
Gastrointestinal symptoms GSRS | Baseline
  GSRS (15 items with values 1-7, total score 1-7 as a mean value of all scores, higher score indicating more severe symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Kaisa Hervonen, PhD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Undecided